CLINICAL TRIAL: NCT00771121
Title: Effect of Moisturizing Creams on Skin Barrier Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ACO Hud Nordic AB (Industry)
Other Study IDs: ACO2008-CT-01
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- new emulsion (Active Comparator)
  Interventions: Drug: urea/lactic acid
- new emulsion placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: urea/lactic acid — new emulsion type
  Arms: new emulsion
Drug: Placebo — only emulsion base
  Arms: new emulsion placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled bilateral study on the effect of moisturizing creams on skin barrier function. The hypothesis is that a new active emulsion has a better influence on skin barrier function comapred to its placebo.

ELIGIBILITY:
Inclusion Criteria:

* Dry skin barrier disorders such as atopic dermatitis or Malassezia eradicated head and neck dermatitis.
* Rough or clinically normal skin on the volar aspect of the forearm.
* Either gender
* Age between 18 and 65 years
* Written Informed Consent

Exclusion Criteria:

* Possible allergy to ingredients in the study medications.
* Use of any concomitant medication that may interfere with the study related activities or assessment of efficacy.
* Any patient related factor suggesting potential poor compliance with study procedures (e.g. psychiatric disorders, history of alcohol or substance abuse).
* Any serious medical condition which, in the opinion of the investigator, may interfere with the evaluation of the results.
* Pregnancy or breast feeding, or patients who plan to become pregnant during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Sophiahemmet, Stockholm, Stockholm County, Sweden